CLINICAL TRIAL: NCT02020187
Title: Aerobic Training in Patients With Congenital Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gitte Hedermann Pedersen, Medical student, Bsc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H2-2013-066
Record Dates: First submitted 2013-11-28; First posted 2013-12-24 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Congenital Myopathy
Keywords: Congenital myopathy; Exercise
MeSH Terms: conditions — Myotonia Congenita; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 10 weeks of home training on a cycle-ergometer. Exercise 30 minutes every other day or at least three times a week.
  Interventions: Other: Exercise on a cycle-ergometer
- Controls (No Intervention): Controls with diagnosed congenital myopathy. Subjects are tested two times on a cycle ergometer. There will be ten weeks between the tests. In between tests the subjects are living life as usual without any interventions.

INTERVENTIONS:
Other: Exercise on a cycle-ergometer — Home training on an ergometer-cycle 30 minutes every other day or at least three times a week. Subject will exercise in a pulse interval corresponding to 70% of their maximal VO2.
  Arms: Exercise

SUMMARY:
Congenital myopathies are clinical and genetic heterogeneous disorders characterized by skeletal muscle weakness. Most patients experience muscle weakness and fatigue throughout their life. However, progression of symptoms is rare. There are no specific treatments for congenital myopathies. Training has been shown to benefit several other muscle diseases with weakness, but the defect in congenital myopathies involves contractile proteins of the sarcomere, why the effect of training is uncertain in these conditions. The investigators will therefore investigate the effect cycle-ergometer training for 30 minutes, three times weakly, for ten weeks in 15 patients with congenital myopathy. Another 5-10 congenital myopathy patients, who do not train, will serve as controls for the trained patients. The study starts and ends with a test day, where efficacy based on VO2max, performance in functional tests and a questionnaire will be assessed.

DETAILED DESCRIPTION:
10 weeks of cycle-ergometer training at home. Intensity at 70% of maximal VO2,max.

ELIGIBILITY:
Inclusion Criteria:

* Danish patients with gene verified congenital myopathy

Exclusion Criteria:

* Patients who are to week to train at a cycle-ergometer for 10 weeks
* Patients who have other health issues, which can disturb the interpretation of the efficacy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy based on VO2,max | 10 weeks
  Difference in VO2,max from baseline to end of intervention.

SECONDARY OUTCOMES:
Level of Creatine Kinase | 10 weeks
  Marker for exercise-induced muscle damage. Taken week 0, 3 and 10.
Intensity in maximal Watt | 10 weeks
  Changes in the maximal intensity (watt) from baseline VO2,max test to after the intervention.
6 minute walk test | 10 weeks
  Changes in the walking distance from baseline to after the intervention.
SF-36 questionnaire | 10 weeks
  Changes in SF-36 questionnaire from baseline to after the intervention.
A timed five-repetitions-sit-to-stand-test | 10 weeks
  Changes in time from baseline to after the intervention.
A timed 14-step-stair-test | 10 weeks
  Changes in time from baseline to after the intervention.
Dynamometry | 10 weeks
  Changes in external force production from baseline to after the intervention. Dynamometry measurements are done at hip flexion, dorsal foot flexion, plantar foot flexion, knee flexion, knee extension and elbow flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte H Pedersen, Bsc Medicine, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Neuromuscular Research Unit, Copenhagen, Denmark

REFERENCES:
- [Derived] Hedermann G, Vissing CR, Heje K, Preisler N, Witting N, Vissing J. Aerobic Training in Patients with Congenital Myopathy. PLoS One. 2016 Jan 11;11(1):e0146036. doi: 10.1371/journal.pone.0146036. eCollection 2016. PMID 26751952